CLINICAL TRIAL: NCT00107913
Title: Phase II Study of Doxil in the Treatment of Patients With Refractory Idiopathic Thrombocytopenic Purpura
Brief Title: Study of Doxil in the Treatment of Patients With Refractory Idiopathic Thrombocytopenic Purpura
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hematology and Oncology Specialists (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOS1
Record Dates: First submitted 2005-04-11; First posted 2005-04-12 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-04

CONDITIONS: Autoimmune Thrombocytopenic Purpura
Keywords: Immune Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — liposomal doxorubicin

INTERVENTIONS:
Drug: Doxil

SUMMARY:
This study is designed to evaluate the efficacy and safety of single agent Doxil in the treatment of patients with refractory ITP (Idiopathic Thrombocytopenic Purpura).

DETAILED DESCRIPTION:
Eligible patients will receive Doxil 20 mg/m2 IV over 1 hour every 2 weeks. Treatment will be continued for 1 course beyond return of the platelet count to normal with a maximum of 18 courses.

ELIGIBILITY:
Inclusion Criteria:

* Thrombocytopenia with bone marrow findings showing normal or increased numbers of megakaryocytes.
* Failure to respond to initial treatment with steroids, IV immune globulin, splenectomy and post splenectomy steroids.
* Platelet count of 30,000 or less.
* Performance status score of 2 or less.
* Adequate organ function: *bilirubin< 2; *AST < 3 times normal; *creatinine < 2.
* No prior treatment with anthracycline or chemically related drugs.

Exclusion Criteria:

* Pregnant or lactating women.
* Presence of a malignancy other than basal cell carcinoma of the skin.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2001-09; Study Completion 2005-04

PRIMARY OUTCOMES:
the primary outcome would be a platelet response, with a return of platelet count to normal

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Cosgriff, MD, Principal Investigator — Hematology and Oncology Specialists
Locations (1):
- Hematology and Oncology Specialists, Metairie, Louisiana, United States